CLINICAL TRIAL: NCT04237558
Title: Laparoscopic Versus Vaginal Hysterectomy in Women With Abnormal Uterine Bleeding Using Bipolar Vessel Sealer in Mansoura University Hospitals: A Randomized Clinical Trial
Brief Title: Laparoscopic Versus Vaginal Hysterectomy in Women With Abnormal Uterine Bleeding Using Bipolar Vessel Sealer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AM1
Record Dates: First submitted 2019-07-26; First posted 2020-01-23 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Uterine Bleeding
Keywords: Vaginal hysterectomy; Laparoscopic hysterectomy
MeSH Terms: conditions — Uterine Hemorrhage | interventions — Hysterectomy, Vaginal

STUDY DESIGN:
Intervention Model Description: comparison between laparoscopic hysterectomy versus non-descent vaginal hysterectomy using bipolar vessel sealers in patients with abnormal uterine bleeding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal hysterectomy (Active Comparator): Removal of uterus through vagina in absence of prolapse
  Interventions: Procedure: Vaginal hysterectomy
- Laparoscopic hysterectomy (Active Comparator): Key hole surgery through small incisions of the abdomen
  Interventions: Procedure: Laparoscopic hysterectomy

INTERVENTIONS:
Procedure: Vaginal hysterectomy — Vaginal hysterectomy by removal of uterus through vagina in absence of prolapse
  Arms: Vaginal hysterectomy
Procedure: Laparoscopic hysterectomy — Laparoscopic hysterectomy through key hole surgery through small incisions of the abdomen
  Arms: Laparoscopic hysterectomy

SUMMARY:
This study will be a randomized clinical trial to evaluate the surgical performance and outcome of total laparoscopic hysterectomy compared to non-descent vaginal hysterectomy ,using bipolar vessel sealer,in cases of abnormal uterine bleeding in Mansoura University Hospital in order to reach the optimum technique for our locality

DETAILED DESCRIPTION:
Hysterectomy is the surgical removal of the uterus. It is the commonest major gynecological surgery, next to caesarean section, with millions of procedures performed annually throughout the world.Approximately 90% of hysterectomies are performed for benign conditions.

Although there are many approaches to hysterectomy, which depend on clinical criteria, certain patients may be eligible to be operated in any of the several available approaches. The optimal route of hysterectomy for a patient will depend on the pathological nature, size and shape of the vagina and uterus, uterine descent, endometriosis and the likelihood of pelvic adhesions, adnexal masses, previous pelvic surgery, available hospital technology, devices and the surgeon's preference.

Approaches to hysterectomy may be broadly categorized into four options: abdominal hysterectomy (AH); vaginal hysterectomy (VH); laparoscopic hysterectomy (LH) where at least some of the operation is conducted laparoscopically and robotic-assisted hysterectomy (RH).Vaginal and laparoscopic procedures are considered "minimally invasive" surgical approaches because they do not require a large abdominal incision and, thus, typically are associated with shortened hospitalization and postoperative recovery times compared with open abdominal hysterectomy.

This study will be a randomized clinical trial to evaluate the surgical performance and outcome of total laparoscopic hysterectomy compared to non-descent vaginal hysterectomy, using bipolar vessel sealer, in cases of abnormal uterine bleeding in order to reach the optimum technique with lower cost to be easily applied to low resource settings.

ELIGIBILITY:
Inclusion Criteria:

* Women assigned for performing hysterectomy for abnormal uterine bleeding due to benign pathology.
* Uterine size by bimanual examination ≤14 weeks gestational size.
* Cases with uterine volumes ≤ 400cm3 will be included in this study.

Exclusion Criteria:

* Patients with BMI > 30kg/m2
* Uteri > 14 weeks gestational size by bimanual examination or volume > 400cm3
* Women with positive pap smear for CIN or endometrial biopsy with atypia or carcinoma.
* Patient with other known body malignancy.
* Patient with other pelvic pathology, endometriosis or pelvic abscesses.
* Patients with abdominal scars.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Duration of operation | From start of surgery up to 24 hours
  Duration of operation

SECONDARY OUTCOMES:
Time of requiring analgesics | Until 24 hours postoperatively
  The time of the first request for analgesics
Number of requiring analgesics | Until 24 hours postoperatively
  The number of requests for analgesics

CONTACTS AND LOCATIONS:
Overall Officials: Amany A Makroum, MSc, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No